CLINICAL TRIAL: NCT01050764
Title: A Feasibility Trial of Post-Transplant Infusion of Allogeneic Regulatory T Cells and Allogeneic Conventional T Cells in Patients With Hematologic Malignancies Undergoing Allogeneic Myeloablative Hematopoietic Cell Transplantation From Haploidentical-Related Donors
Brief Title: Haploidentical Allogeneic Transplant With Post-transplant Infusion of Regulatory T-cells
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Safety
Sponsor: Everett Meyer (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor-Investigator, Everett Meyer, Assistant Professor of Medicine (Blood and Marrow Transplantation), Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-15919; BMT204 (Other: OnCore); SU-03312009-2059 (Other: Stanford University)
Record Dates: First submitted 2010-01-11; First posted 2010-01-15 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Leukemia, Acute; Chronic Myelogenous Leukemia (CML); Myelodysplastic Syndrome (MDS); Non-Hodgkin Lymphoma (NHL); Chronic Lymphocytic Leukemia (CLL); Acute Myelogenous Leukemia (AML); Acute Lymphoblastic Leukemia (ALL)
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Melphalan; Thiotepa; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- T-reg Cell Infusion after Allogeneic Stem Cell Transplant (Experimental)
  Interventions: Drug: Regulatory T-cells; Drug: Conventional T-cells; Drug: Melphalan; Drug: Thiotepa; Device: Fludarabine; Drug: Anti-thymocyte globulin, rabbit; Drug: CliniMACS CD34 Reagent System

INTERVENTIONS:
Drug: Regulatory T-cells — To ameliorate the impaired immune recovery and address the significant relapse incidence in the haploidentical setting. Cells will be selected by a tandem selection process and infused on day +14. These are the enriched but naturally-occurring regulatory T cells. Possible dose cohorts and levels are:
  Cohort 1
  * T-reg: 1 x 10e5/kg
  * T-con: 3 x10e5/kg
  Cohort 2
  * T-reg: 3 x 10e5/kg
  * T-con: 1 x 10e6/kg
  Cohort 3
  * T-reg: 1 x 10e6/kg
  * T-con: 3 x 10e6/kg
  Cohort 4
  * T-reg: 3 x 10e6/kg
  * T-con: 1 x 10e7/kg
  Other Names: T-reg cells
Drug: Conventional T-cells — These are conventional (unselected) donor T-cells. Cell dosage of the infusion will be based on the CD3+ cell content and infused on day +16.
  Other Names: T-con cells
Drug: Melphalan — Anti-cancer chemotherapy drug administered IV at 140 mg/m² on Day -8 prior to HSCT (a component of the conditioning regiment prior to infusion of cells)
  Other Names: L-PAM; L-Sarcolysin; Phenylalanine Mustard
Drug: Thiotepa — Anti-cancer chemotherapy drug administered IV at 10 mg/kg on Day -7 prior to HSCT (a component of the conditioning regiment prior to infusion of cells)
  Other Names: thiophosphamide; TESPA; TSPA
Device: Fludarabine — Anti-cancer chemotherapy drug administered IV at 160mg/m² on Days -6; -5; -4; and -3 prior to HSCT (a component of the conditioning regiment prior to infusion of cells
  Other Names: Fludarabine phosphate; Fludarabine 5'-monophosphate; FAMP; Fludara
Drug: Anti-thymocyte globulin, rabbit — Rabbit-derived antibodies against human T-cells used as transplant rejection prophylaxis. Administered at 6 mg/kg IV on Days -6; -5; -4; and -3 prior to HSCT
  Other Names: Thymoglobulin; rATG
Drug: CliniMACS CD34 Reagent System — An in vitro medical device system that uses antibodies conjugated to magnetic beads to select and enrich for CD34+ blood stem cells from the allogeneic donor apheresis product prior to HSCT, while removing other cells that can cause GvHD. CD34+ cell dosage will be based on the participant's body weight.

SUMMARY:
Patients with hematologic malignancies will receive myeloablative chemotherapy followed by stem cell rescue with bone marrow or hematopoietic peripheral blood stem cells collected by apheresis from a filgrastim- (G-CSF)-mobilized haploidentical related-donor, ie, hematopoietic peripheral blood stem cell transplant (HSCT).

DETAILED DESCRIPTION:
This is dose-escalation study intended to evaluate the use of classification determinant 15-positive (CD15+), CD4+, CD127dim, and FoxP3+ regulatory T-cells (T-reg cells) supplemented by conventional T-cells (T-con cells), to enhance the efficacy of allogeneic (CliniMACS CD34+ selected) hematopoietic stem cell transplantation (allo-HSCT), in the setting of leukemia, lymphoma, and myelodysplastic syndrome (MDS). This study investigates amelioration of the impaired immune recovery and address the significant relapse incidence in the haploidentical HSCT setting.

Pre-transplant myeloablative conditioning will be melphalan; thiotepa; fludarabine and rabbit antithymocyte globulin (rATG).

Stem cell rescue will be with CD34+ selected cells. The rescue infusion will be supplemented with infusions of regulatory T-cells (T-reg) and conventional T-cells (T-con) from the same donor collection, on Treatment Days 14 and 16 respectively. CD34+ cell infusion day is Treatment Day 0.

T-reg cells are those cells enriched by immunomagnetic selection of CD25+ cells, and further purified by flow cytometric cell sorting for the CD15+, CD4+, CD127dim, FoxP3+ cell population. These cells are an enriched but naturally-occurring T-cell population.

T-con cells are unseparated/unfractionated cells, ie, as collected by the peripheral blood stem cells apheresis procedure.

Post-transplant follow-up is for 5 years.

ELIGIBILITY:
Inclusion Criteria

RECIPIENT

* Histopathologically-confirmed:
* Acute leukemia (in first remission with poor risk factors and molecular prognosis)
* Acute myelogenous leukemia (AML) with -5,-7, t (6;9), tri8, -11
* Acute lymphoblastic leukemia (ALL) with Ph+ t (9;22), t (4;22), (q34;q11)
* Acute leukemia with refractory disease or > Complete Remission (CR) 1
* Chronic myelogenous leukemia (CML) (accelerated, blast or second chronic phase)
* Myelodysplastic syndrome (in high and high intermediate risk categories)
* Non-Hodgkin's lymphoma (NHL) with poor risk features and not suitable for autologous transplantation
* Refractory Chronic lymphocytic leukemia (CLL)
* At least 21 days from the end of most recent prior therapy to start of the transplant conditioning regimen
* Must be < 60 years old at time of registration.
* Karnofsky Performance Status (KPS) > 70%

Must have related donor who is:

* Genotypically human leukocyte antigen (HLA) -A, B,C and DR beta 1 (DRB1), DQ loci haploidentical to the recipient (but differing for 2 to 3 HLA alleles on the unshared haplotype in the graft-versus-host disease (GvHD) direction)
* No HLA-matched sibling or matched-unrelated donor is identified.
* Adequate cardiac and pulmonary function (left ventricular ejection fraction (LVEF) > 45%, diffusing capacity of the lungs for carbon monoxide (DLCO) >50% corrected for hemoglobin)
* Serum creatinine < 1.5 mg/dL OR Creatinine clearance > 50 mL/min for those above serum creatinine at least 1.5 mg/dL
* Serum bilirubin < 2.0 mg/dL
* Alanine transaminase (ALT) < 2x upper normal limit (ULN) (unless secondary to disease)
* No prior myeloablative therapy or hematopoietic cell transplantation

DONOR:

* Age ≤ 70 years
* Weight ≥ 25 kg.
* Medical history and physical examination confirm good health status as defined by institutional standards
* Seronegative for HIV Ag within 30 days of apheresis collection for:
* Hepatitis B surface antigen (sAg) or polymerase chain reaction (PCR) +
* Hepatitis C ab or PCR+
* Genotypically haploidentical as determined by HLA typing
* Female donors (child-bearing potential) must have a negative serum or urine beta-human chorionic gonadotropin (HCG) test within 3 weeks of mobilization
* Capable of undergoing leukapheresis
* Has adequate venous access
* Willing to undergo insertion of a central catheter if leukapheresis via peripheral vein is inadequate
* Capable of agreeing to second donation of peripheral blood progenitor cell (PBPC) (or a bone marrow harvest) should the patient fail to demonstrate sustained engraftment following the transplant
* Institutional review board (IRB)-approved consent form signed by donor or legal guardian > 18 years of age

Donor Selection in the priority order:

* Recipient's biological mother preferred, if available
* Other available haploidentical donors will be selected based upon the presence of natural killer (NK) alloreactivity between donor and recipient by high-resolution HLA typing of the C locus. An NK-alloreactive donor will be preferentially chosen. Recipients lacking a killer immunoglobulin-like receptor (KIR)-ligand present in the donor along with the corresponding KIR defines "NK alloreactivity".
* If more than one NK-alloreactive donor is available, preference is to cytomegalovirus (CMV)-seronegative donor

Exclusion Criteria

RECIPIENT:

* Suitable candidate for autologous transplantation or allogeneic transplantation with an available matched-related or matched-unrelated donor
* Seropositive for:
* HIV ab
* Hepatitis B sAg or PCR+
* Hepatitis C ab or PCR+
* History of invasive Aspergillosis
* Any active, uncontrolled bacterial, viral or fungal infection
* Uncontrolled central nervous system (CNS) disease involvement
* Lactating female

DONOR:

* Evidence of active infection or viral hepatitis
* Factors of increased risk for complications from leukapheresis or granulocyte-colony stimulating factor (G-CSF) therapy
* Lactating female
* HIV-positive

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett H Meyer, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Allogeneic T-Cell Infusion After Stem Cell Transplant (SCT): Allogeneic, haploidentical hematopoietic stem cell transplant (allo-HSCT) of bone marrow and/or peripheral blood stem cells, followed by infusion of regulatory T-cells (T-reg) plus conventional CD4 and CD8 T-cells (T-con)
Period: Overall Study
Arm/Group | Allogeneic T-Cell Infusion After Stem Cell Transplant (SCT)
Started | 10
Received HSCT Graft | 8
Received Infusion of T-reg Cells | 7
Received Infusion of T-con Cells | 7
Completed | 7
Not Completed | 3
Not completed — Death, before HSCT | 1
Not completed — Donor mobilization failure, death | 1
Not completed — Death after HSCT, before T-cell infusion | 1

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic T-Cell Infusion After Stem Cell Transplant (SCT)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose (MTD) of Regulatory and Conventional T-cells
Description: The maximum-tolerated dose (MTD) was to be determined based on the safety and feasibility observed for a pre-determined set of cellular dose level combinations of regulatory T-cells (T-reg) and conventional T-cells (T-con).
Time Frame: 30 days after HSCT infusion
Population: Includes all participants that received HSCT
Measure: Number; unit: cells/kg
Arm/Group | Allogeneic T-Cell Infusion After Stem Cell Transplant (SCT)
Number analyzed (Participants) | 8
cells/kg | NA — GvHD was within parameters to continue, but the study was terminated due to poor outcomes prior to sufficient accrual to set the MTD, even at the only dose level tested (1x10e5/kg T-reg cells + 1x10e5/kg T-con cells). Primary outcome result is null.

2. Secondary Outcome: Acute Graft-versus-Host-Disease (aGvHD)
Description: The primary outcome was incidence of grade 3 or 4 acute graft-vs-host-disease (aGvHD), reported as the number of participants developing grade 3 or 4 aGvHD.
Time Frame: 1 year
Population: Population of participants that received HSCT and T-reg plus T-con
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic T-Cell Infusion After Stem Cell Transplant (SCT)
Number analyzed (Participants) | 7
Participants | 1

3. Secondary Outcome: Overall Survival (OS), 1 Year
Description: Assessed as subjects remaining alive 12 months after CD34+ cell infusion (ie, excludes death due to any cause)
Time Frame: 1 year
Population: Population of participants that received HSCT and T-reg plus T-con
Measure: Number; unit: Participants
Arm/Group | Allogeneic T-Cell Infusion After Stem Cell Transplant (SCT)
Number analyzed (Participants) | 7
Participants | 2

4. Secondary Outcome: Median Overall Survival (OS)
Description: Reported as the median overall survival (OS) in months from infusion of the hematopoietic stem cells (HSCT)
Time Frame: 25 months
Population: Population of participants that received HSCT and T-reg plus T-con
Measure: Median (Standard Deviation); unit: months
Arm/Group | Allogeneic T-Cell Infusion After Stem Cell Transplant (SCT)
Number analyzed (Participants) | 7
months | 3.7 (10)

5. Secondary Outcome: To Measure the Incidence and Severity of Acute and Chronic GvHD
Description: Population of participants that received HSCT and T-reg plus T-con, and developed actue, chronic, or any graft vs host disease (GvHD)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic T-Cell Infusion After Stem Cell Transplant (SCT)
Number analyzed (Participants) | 7
Participants
  Acute GvHD | 1
  Chronic GvHD | 2
  Any GvHD (actue + chronic) | 3

6. Secondary Outcome: Serious Infections
Description: Serious infections are reported as the number of participants experienced serious infections.
Time Frame: 1 year
Population: Population of participants that received HSCT and T-reg plus T-con
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic T-Cell Infusion After Stem Cell Transplant (SCT)
Number analyzed (Participants) | 7
Participants | 6

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse events are only reported for those participants that received the allogeneic T-cell Infusion after the stem cell transplant (SCT). Those that did not receive the SCT, or received only the SCT but the T-cell infusion, are not included except in the all-cause mortality data.
Arm/Group | Allogeneic T-Cell Infusion After Stem Cell Transplant (SCT)
All-Cause Mortality (participants affected / at risk) | 9/9
Serious Adverse Events (participants affected / at risk) | 7/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic T-Cell Infusion After Stem Cell Transplant (SCT) (N=7)
Acute graft vs host disease (GvHD) (Immune system disorders) | 3 (3) — Liver, gut, skin
Acute renal failure (Renal and urinary disorders) | 2 (2)
Adenoviral infection (Infections and infestations) | 4 (4)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bacteremia (Infections and infestations) | 3 (3)
Cardiorespiratory failure (General disorders) | 1 (1)
Death (General disorders) | 1 (1) — Not otherwise specified
Diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypocellular marrow (Blood and lymphatic system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Progressive disease / relapse / recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic T-Cell Infusion After Stem Cell Transplant (SCT) (N=7)
Acute graft vs host disease (aGvHD), gut (Immune system disorders) | 1 (1)
aGvHD, liver (Immune system disorders) | 1 (1)
aGvHD, skin (Immune system disorders) | 3 (3)
Neutropenic fever (Blood and lymphatic system disorders) | 2 (2)
Hemorrhagic cystitis (Gastrointestinal disorders) | 2 (2)
Mucositis (Gastrointestinal disorders) | 2 (2)
Edema, lower extremity (General disorders) | 1 (1)
Pain, abdominal (General disorders) | 1 (1)
Infection (Infections and infestations) | 7 (15)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No